CLINICAL TRIAL: NCT03153982
Title: Pharmacodynamic Effects and Predictive Biomarkers of Janus Kinases (JAK)/Signal Transducer and Activator of Transcription (STAT) Inhibition With Ruxolitinib in Operable Head and Neck Cancer: a Window Trial
Brief Title: Ruxolitinib in Operable Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16201; NCI-2017-02304 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: JAK/STAT inhibition; Biomarkers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant Ruxolitinib (Experimental): Participants will take 15 mg or 20 mg of ruxolitinib by mouth twice daily for up to 4 weeks during the pre-operative window for 14-21 days, or up to 28 days for delays in planned surgery. Dose will be assigned based on participant platelet count at baseline. The last dose will be taken the morning of planned surgery. Ruxolitinib will be dispensed in 5 mg tablets. Participants will either take three tables (15 mg) in the morning and evening, or four tablets in the morning and evening (20 mg). Participants will be asked to fill out a drug diary indicating when doses of study drug are taken and any side effects they experience.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Given orally
  Other Names: Jakafi

SUMMARY:
The purpose of this study is to assess the safety and efficacy of ruxolitinib in patients with operable Head and neck squamous cell carcinoma (HNSCC) who are planned for definitive surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify baseline and/or pharmacodynamic biomarkers of response to ruxolitinib, based upon association with quantitative change in tumor size following 14-21 days of neoadjuvant ruxolitinib in patients with operable HNSCC as determined by quantitative change in Tumor size.

SECONDARY OBJECTIVES:

I. To describe the tolerability of brief neoadjuvant exposure to ruxolitinib II. To assess the effect of ruxolitinib on the tumoral Ki-67 proliferation index III. To evaluate additional candidate biomarkers of ruxolitinib response or resistance in HNSCC patients as determined by quantitative change in Tumor size,

OUTLINE:

Participants will be assigned neoadjuvant ruxolitinib based on participant platelet counts at baseline. Participants with a platelet count of 200,000 or greater will take 20 mg twice daily and participants with a platelet count between 150,000 and 200,000 will take 15 mg twice daily. Participants may continue treatment for up to 4 weeks from the time of study entry to time of planned standard of care surgery for cancer. Participants will be followed up for 12-weeks post-operation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, primary or recurrent, head and neck squamous cell carcinoma, including variants. Patients must have at least one measureable lesion in accordance with RECIST 1.1 (tumor diameter ≥ 1 cm; short-axis lymph node diameter ≥ 1.5 cm) OR by caliper measurement (tumor diameter ≥ 1 cm). Any diagnostic pretreatment biopsy sample is acceptable including fine needle aspiration (FNA).
2. Primary tumors of any head and neck (oral cavity, oropharynx, hypopharynx, or larynx) site will be included.
3. Surgical resection of head and neck must be planned, either as primary treatment or salvage. Patients must have submitted adequate pretreatment archival or fresh tissue.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (See Appendix 1).
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (sensitivity ≤ 25 human chorionic gonadotropin (HCG) IU/L) within 4 weeks prior to registration and will be repeated within 72 hours prior to the start of study drug administration.
7. Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 12 weeks after study drug is stopped. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
8. Adequate hematologic, renal and hepatic function, as defined by:

   1. Absolute neutrophil count (ANC) ≥ 1,500/ul, platelets ≥ 150,000/ul.
   2. Creatinine ≤ 1.5 x institutional upper limit of normal (ULN).
   3. Bilirubin ≤ 1.5 x ULN, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x ULN.
9. Have signed written informed consent

Exclusion Criteria:

1. Subjects who fail to meet the above criteria.
2. Prior therapy for head and neck cancer is allowed, and the number of treatments is not limited. However, any systemic therapy should have been completed at least 30 days prior to study enrollment. Any radiation to the head and neck should have been completed at least 30 days prior to study enrollment. Palliative radiation outside of the head and neck does not require a washout.
3. Pregnancy or breastfeeding. Women (patients or partners of male patients) of childbearing potential (WOCBP) must practice acceptable methods of birth control to prevent pregnancy. All WOCBP must have a negative pregnancy test within 4 weeks prior to registration, and this must be repeated within 72 hours prior to first receiving ruxolitinib. If the pregnancy test is positive, the patient must not receive ruxolitinib and must not be enrolled in the study.
4. Any unresolved chronic toxicity ≥ grade 2 from previous anticancer therapy (except alopecia and anemia), according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
5. Current active infection requiring systemic antibiotic or antifungal therapy.
6. Acute hepatitis or known HIV.
7. Treatment with a non-approved or investigational drug within 30 days prior to Day 1 of study treatment.
8. New York Heart Association (NYHA) Class III or IV heart disease.
9. History of thromboembolic event or other condition currently requiring anticoagulation with warfarin (coumadin). Patients who are treated with low molecular weight heparin or fondaparinux are eligible.
10. History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease, diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies, or ongoing or recent (≤ 3 months) significant gastrointestinal bleeding
11. Concomitant Medications, any of the following should be considered for exclusion: Strong CYP3A4 inhibitors: (Patients must discontinue drug 7 days prior to starting ruxolitinib), including but not limited to boceprevir, clarithromycin, conivaptan, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, or voriconazole. In addition, patients will be instructed to avoid grapefruit or grapefruit juice, starfruit, or seville oranges.
12. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Ryan, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qureshy Z, Li H, Zeng Y, Rivera J, Cheng N, Peterson CN, Kim MO, Ryan WR, Ha PK, Bauman JE, Wang SJ, Long SR, Johnson DE, Grandis JR. STAT3 Activation as a Predictive Biomarker for Ruxolitinib Response in Head and Neck Cancer. Clin Cancer Res. 2022 Nov 1;28(21):4737-4746. doi: 10.1158/1078-0432.CCR-22-0744. PMID 35929989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Ruxolitinib
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Ruxolitinib
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 1
  50-59 years old | 6
  60-69 years old | 3
  70-79 years old | 5
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportional Percent Change in Tumor Size by Group
Description: Measured clinical ruxolitinib response of quantitative change in tumor size measured as a proportional percent (range -100% to +100%) from baseline to day 14-21 by group.
Time Frame: Up to 4 weeks
Population: Data not collected
Arm/Group | Neoadjuvant Ruxolitinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: The number of participants with treatment-related adverse events, defined as definite, probable or possibly related to the study intervention and classified according to NCI CTCAE version 4 will be reported.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Ruxolitinib
Number analyzed (Participants) | 16
Participants | 1

3. Secondary Outcome: Number of Participants With Documented Surgical Complications
Description: The number of participants with documented surgical complications will be reported.
Time Frame: Up to 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Ruxolitinib
Number analyzed (Participants) | 16
Participants | 0

4. Secondary Outcome: Median Length of Hospital Stay
Description: The median length of hospital stay following the standard of care, surgical procedure will be reported.
Time Frame: Up to 12 weeks
Population: Hospital stay length data not collected
Arm/Group | Neoadjuvant Ruxolitinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Change in Ki-67 Proliferative Index Value
Description: A high Ki-67 proliferation index means many cells are dividing quickly and that the cancer is likely to grow and spread. A Ki-67 proliferation index over 30% is typically considered high. The Ki-67 proliferative index will be measured at baseline and post-treatment tumor tissue.
Time Frame: Up to 12 weeks
Population: Ki-67 proliferative index data not collected
Arm/Group | Neoadjuvant Ruxolitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Neoadjuvant Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Ruxolitinib (N=16)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Ruxolitinib (N=16)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Non-cardiac chest pain (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Investigations) | 1 (1)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Tissue sloughing off tumor (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed earlier than expected due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT03153982/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03153982/ICF_001.pdf